CLINICAL TRIAL: NCT04862104
Title: The Effect of Discharge Training on Surgical Recovery in Oncology Patients: A Randomized Control Trial
Brief Title: The Effect of Discharge Training on Surgical Recovery in Oncology Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Ezgi Arslan, Research Assistant, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Surgical Recovery
Record Dates: First submitted 2021-04-23; First posted 2021-04-27 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Surgery--Complications; Nursing Caries
Keywords: Surgical recovery; Discharge Training; Follow-up; Nursing

STUDY DESIGN:
Intervention Model Description: Following recruitment, patient who underwent oncological surgery were divided into a study and a control group by randomization (1:1 randomization)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Discharge Training) (Experimental): In addition to the general care provided by health professionals, the study group received discharge training created according to the Nursing Interventions Classification.
  Interventions: Behavioral: Intervention group
- Control group (Usual Care) (No Intervention): The control group continued to receive the routine care

INTERVENTIONS:
Behavioral: Intervention group — In addition to the routine care they received, the patients in the intervention groups were given discharge training developed in the pre-discharge period. Discharge training consisted of a verbal and written information booklet containing instructions for the patient and the patient's caregiver on pain management, nutrition management, incision site care, strengthening self-care, returning to daily life activities, and colostomy care. Discharge training was given in the service after evaluating the surgical recovery status of the patient before discharge. The average duration of each training was 30-45 minutes. The patients were evaluated in terms of surgical recovery by calling by phone 2 weeks after discharge, 4 weeks and 8 weeks later. The developed education booklet was given to the patient and it was ensured that he could benefit from the information at home.
  Arms: Intervention group (Discharge Training)

SUMMARY:
A randomized control trial was made to examine the effect of discharge training developed using Nursing Interventions Classification on surgical recovery in patient who underwent oncological surgery.

DETAILED DESCRIPTION:
The concept of surgical recovery is defined as "starting activities aimed at maintaining daily life, health and well-being after surgery" and delay in surgical recovery "increasing the number of days after surgery required to start activities aimed at maintaining daily life, health and well-being after surgery". Problems such as fatigue, pain, incisional surgical site infection, loss of appetite, which are common in patients in the postoperative period, are symptoms associated with delayed surgical recovery. In addition to these symptoms, the presence of conditions such as delayed return to home / work activities need for self-care, nausea, anorexia, pain, and difficulty in moving indicate that surgical recovery is interrupted. It has been reported that delay in surgical recovery is common after surgeries such as gastrostomy, colectomy, and exploratory laparotomy.

Patients who have undergone gastric or colorectal cancer surgery should receive discharge training before returning to social life and business life. Nurses should determine the problems they may experience at home in patients who have undergone surgeries such as gastrostomy, colectomy, and exploratory laparotomy, where delay in surgical recovery is frequently reported, plan and apply discharge training for these problems, and monitor patients in terms of surgical recovery processes at home. It has been reported that this way, the surgical recovery process can be supported and delays in surgical recovery can be prevented.

This study was conducted to determine the effect of a discharge training developed using the Nursing Interventions Classification on surgical recovery in patients undergoing oncologic surgery.

It was tested the hypotheses that there was no difference between the post-intervention intervention and control groups in terms of the surgical recovery score averages in patients who had undergone oncologic surgery were tested.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18 and 75
* Stomach or colorectal surgery
* Volunteering to participate in research
* Understanding and speaking Turkish
* Having a telephone that can be reached by him or his caregiver

Exclusion Criteria:

* Responding to less than 75% of phone calls
* Not having cognitive functions in place
* Having a hearing problem
* Not having a relative to answer in case he / she cannot answer the phone
* Having complications during hospitalization (ileus, septic shock, herniation)
* Having a history of chemotherapy / radiotherapy in the last two months
* To receive chemotherapy / radiotherapy within two months after surgery
* Complications developed during surgery
* To be transferred to the intensive care unit after surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-12-27 (Actual)

PRIMARY OUTCOMES:
The surgical recovery score averages in patients | before discharge in the postoperative days
  assessed using the Patient Evaluation Form, nine defining features of the diagnosis of "delayed surgical recovery" defined in NANDA-I (delaying starting activities at home / work, understanding that more time is required for recovery/ recovery, need for assistance in self-care practices, evidence indicating impaired surgical site presence (discharge, swelling, redness, pain, presence of one of the bleeding in the area mild; the presence of all will be marked as severe distress), loss of appetite with nausea, loss of appetite without nausea, difficulty in moving around, pain or discomfort, fatigue) It contains questions.
  The patient evaluation form was created using the Nursing Outcomes Classification of the five-point Likert-type scale measuring the severity of descriptive features. The expression "severely distressed" was "1 point"; The expression "significantly distressed" was evaluated as "2 points", "moderately distressed" as "3 points", "mildly distressed" as "4 points", and "no
The surgical recovery status after intervention | In the second weeks after discharge
  assessed using the Patient Evaluation Form. The form is composed of nine items. The form is The expression "severely distressed" was "1 point"; The expression "significantly distressed" was evaluated as "2 points", "moderately distressed" as "3 points", "mildly distressed" as "4 points", and "no distress" as "5 points". The patient can get a minimum of nine and a maximum of 45 points. As the score for each evaluation question increased, the improvement was evaluated as positive. It was applied by telephone in the second week after discharge.
The surgical recovery status after intervention | In the fourth weeks after discharge
  assessed using the Patient Evaluation Form. The form is composed of nine items. The form is The expression "severely distressed" was "1 point"; The expression "significantly distressed" was evaluated as "2 points", "moderately distressed" as "3 points", "mildly distressed" as "4 points", and "no distress" as "5 points". The patient can get a minimum of nine and a maximum of 45 points. As the score for each evaluation question increased, the improvement was evaluated as positive. It was applied by telephone in the fourth week after discharge.
The surgical recovery status after intervention | In the eighth weeks after discharge
  assessed using the Patient Evaluation Form. The form is composed of nine items. The form is The expression "severely distressed" was "1 point"; The expression "significantly distressed" was evaluated as "2 points", "moderately distressed" as "3 points", "mildly distressed" as "4 points", and "no distress" as "5 points". The patient can get a minimum of nine and a maximum of 45 points. As the score for each evaluation question increased, the improvement was evaluated as positive. It was applied by telephone in the eighth week after discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Ezgi Arslan, PhD Student, Principal Investigator — Aydın Adnan Menderes University, Faculty of Nursing, Surgical Nursing Department
Locations (1):
- Aydın Adnan Menderes University, Aydin, Efeler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: CSR
Time Frame: 6 months after publication
Access Criteria: Relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.

REFERENCES:
- [Derived] Arslan E, Gezer N. The effect of discharge training developed based on nursing interventions classification (NIC) on surgical recovery in oncology patients: Randomized controlled trial - A pilot study. Nurs Open. 2023 Feb;10(2):1151-1162. doi: 10.1002/nop2.1555. Epub 2022 Dec 25. PMID 36567264